CLINICAL TRIAL: NCT03969485
Title: Non-Randomized, Open-label, Blinded Evaluator Study Characterizing Effectiveness of Hybrid Fractional Laser for the Treatment of Off Face Body Skin Quality
Brief Title: Hybrid Fractional Laser for Treatment of Off Face Body Skin Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HALOCIP002
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid Fractional Laser (Experimental): Hybrid Fractional Laser Treatment
  Interventions: Device: Hybrid Fractional Laser

INTERVENTIONS:
Device: Hybrid Fractional Laser — Hybrid Fractional Laser Device
  Other Names: HALO

SUMMARY:
To demonstrate effectiveness of hybrid fractional laser for the treatment of poor skin quality on the decolletage, back of the hands and lower legs

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male/female subjects between 40 to 65 years of age inclusive
2. Fitzpatrick skin type I-III
3. Non-smokers or have not smoked (including vaping) within the past 14 days from the screening visit
4. Has poor skin texture
5. Has mild thin skin
6. Has some level of dyschromia on the treatment area as assessed by the Investigator
7. Can read, understand and sign informed consent form (English only)
8. Has indicated willingness to participate in the study by signing an informed consent form
9. Agrees to adhere to the treatment and follow-up schedule and post treatment care instructions

Exclusion Criteria:

1. Fitzpatrick skin type IV-VI
2. Has tanned within the past 30 days or is unable or unlikely to refrain from tanning, including the use of tanning booths, tanning spray or cream
3. Has tattoos, dysplastic nevi on the treatment area
4. Is pregnant and/or lactating
5. History or current photosensitivity
6. History or current use of medication with photosensitizing properties within past 6 months
7. History or current of chronic reoccurring skin disease or disorder affecting treatment area
8. History or current cancer of any type
9. Has signs of actinic bronzing
10. Has open lacerations, and abrasions on the treatment area
11. History of keloid formation, or hypertrophic scar formation, or poor wound healing
12. History of bleeding disorder, or is currently taking anticoagulation medications
13. Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, which might be aggravated as a result of treatment
14. Has participated in any clinical trial involving an investigational drug, device or cosmetic product or procedure within the past 30 days
15. The investigator feels that for any reason the subject is not eligible to participate in the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Photography | 3 months
  Evaluate improvement in photography using Physicians Global Assessment Scale (0-4) where 0 is no change and 4 is very significant improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- New Jersey Clinical Research Center, Montclair, New Jersey, United States